CLINICAL TRIAL: NCT06359314
Title: Positive Emotion Regulation Intervention for Benzodiazepine Receptor Agonist Deprescribing in Older Adults: Anxiety Lowering and Deprescribing Through Emotion Regulation (ALDER)
Brief Title: Anxiety Lowering and Deprescribing Through Emotion Regulation
Acronym: ALDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Elizabeth Addington, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00219362
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Benzodiazepine Dependence; Anxiety Disorders; Sleep Disturbance
Keywords: Benzodiazepine receptor agonists; Positive emotion; Sleep disturbance; Anxiety; Coping; Stress
MeSH Terms: conditions — Anxiety Disorders; Parasomnias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will go through a 5-week online self-guided positive emotion skills course.
  Interventions: Behavioral: ALDER

INTERVENTIONS:
Behavioral: ALDER — The ALDER skills are delivered over approximately 5 weeks. A week consists of learning at least one skill and then applying that skill(s) in daily home practice throughout the week. Skill lessons and daily home practice exercises are housed on the ALDER website. Participants have the option to share their home practice responses with fellow participants by posting them to the discussion board, where they can like and comment on each other's posts.

SUMMARY:
The goal of this clinical trial is to test ALDER (Anxiety Lowering and Deprescribing through Emotion Regulation), an online self-guided positive emotion intervention, in patients over the age of 65 who are candidates for benzodiazepine receptor agonist (BZRA, commonly called benzos, or z-drugs) deprescribing. The main questions it aims to answer are:

* Is ALDER relevant to and satisfactory for older adult BZRA users?
* Does ALDER help to increase positive emotions and decrease anxiety, trouble sleeping, and use of BZRA medications?

Participants will complete the 5-week online self-guided ALDER intervention as well as two survey assessments, one before the intervention and one after.

DETAILED DESCRIPTION:
ALDER (Anxiety Lowering and Deprescribing through Emotion Regulation) is a pilot trial of an online positive emotion intervention for adults age 65 and over who are candidates for benzodiazepine receptor agonist (BZRA) deprescribing. The ALDER intervention is 5 weeks long and involves weekly self-guided positive emotion skill lessons and daily skill practice exercises, both housed on the ALDER website.

Up to n=40 patients over the age of 65 will be recruited from Northwestern Medicine Primary Care clinics. To participate, patients must have (1) a BZRA prescription from Northwestern Medicine Primary Care within the past year, (2) at least 1 NM Primary Care visit in the past year, and (3) take a BZRA at least twice a week. Participants will complete survey assessments via REDCap before and after they go through the ALDER intervention. All study activities will take place online.

Feasibility, acceptability, and adoption of the ALDER program will be assessed using enrollment and retention rates, website user data, and measures of relevance and satisfaction in the post-intervention assessment. Patient reported outcomes such as anxiety, sleep and positive affect will be measured both pre- and post-intervention and rate of BZRA usage will be extracted from participant medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and over.
* ≥1 NM Internal Medicine clinic visit within the past year.
* BZRA prescribed by NM primary care within the past year.
* Takes BZRA at least twice a week.
* Daily access to internet-connected device.
* Ability to read and speak English.

Exclusion Criteria:

* Dementia, seizure, or REM sleep disorder diagnosis.
* In hospice care.
* No daily internet access.
* Cannot speak and read English.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Addington, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Northwestern Medicine using electronic messages.
Pre-assignment Details: Participants who met all eligibility requirements and provided informed consent were given access to the web-based intervention.
Period: Overall Study
Arm/Group | Intervention
Started | 33
Completed | 16
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Comorbidities [Mean (Standard Deviation); unit: number of comorbid chronic health condit] — Self-reported health conditions
  number of comorbid chronic health condit | 2.35 (1.6)
Reasons for BZRA use [Count of Participants; unit: Participants] — Self-reported reason(s) for using benzodiazepine receptor agonist (BZRA) medication(s)
  Participants
    Anxiety or stress only | 9
    Sleep only | 17
    Both anxiety/stress and sleep | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention
Description: Measured by enrollment rate (# consented/# eligible) and retention rate (# of complete post-intervention assessments/# consented).
Time Frame: Measured post-intervention (7-weeks).
Population: n=49 were eligible; n=33 consented; n=16 were retained at post-intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 49
Percentage of participants
  Enrollment rate | 67
  Retention rate: number analyzed (Participants) | 33
  Retention rate | 48

2. Primary Outcome: Acceptability of Intervention
Description: Measured during the post-intervention assessment using the Acceptability of Intervention Measure to evaluate relevance of and satisfaction with the ALDER intervention. Examples of survey items include "ALDER meets my approval" and "I like ALDER." The final score is an average of the scores from 4 items. Maximum score is 5, minimum score is 1. Higher scores indicate greater acceptability.
Time Frame: Measured post-intervention (7-weeks).
Population: n=16 provided data at post-intervention
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Intervention
Number analyzed (Participants) | 16
Scores on a Scale | 3.72 (1.1)

3. Primary Outcome: Adoption of Intervention
Description: Measured via usage metrics from the BrightOutcome intervention platform (e.g., mean number of skills accessed).
Time Frame: Measured post-intervention (7-weeks).
Measure: Mean (Standard Deviation); unit: number of skills used (min 0, max 8)
Arm/Group | Intervention
Number analyzed (Participants) | 33
number of skills used (min 0, max 8) | 4 (3.5)

4. Secondary Outcome: Patient Benzodiazepine Receptor Agonist (BZRA) Use
Description: Three questions asking patients which medication they use, their frequency of use (times per week), and their reason for use (anxiety, stress, sleep, other).
Time Frame: Measured at baseline (pre-intervention) and post-intervention (7-weeks).
Measure: Median (Full Range); unit: days per week
Arm/Group | Intervention
Number analyzed (Participants) | 33
days per week
  Baseline BZRA usage | 6 [1 to 7]
  Post-intervention BZRA usage | 5 [2 to 7]

5. Secondary Outcome: Patient-reported Sleep Disturbance
Description: Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0 - Sleep Disturbance computer adaptive test, which assesses self-reported perceptions of sleep quality, depth, and restoration within the past 7 days, including difficulty falling asleep and staying asleep and sleep satisfaction. Higher scores indicate higher levels of sleep disturbance. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Measured at baseline (pre-intervention) and post-intervention (7-weeks).
Population: n=16 were retained at post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention
Number analyzed (Participants) | 33
T-score
  Baseline sleep disturbance | 54.39 (8.01)
  Post-intervention sleep disturbance: number analyzed (Participants) | 16
  Post-intervention sleep disturbance | 52.79 (10.11)

6. Secondary Outcome: Patient-reported Anxiety
Description: Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0 - Anxiety computer adaptive test, which assesses self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Higher scores indicate higher levels of anxiety. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Measured at baseline (pre-intervention) and post-intervention (7-weeks).
Population: n=16 were retained at post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention
Number analyzed (Participants) | 33
T-score
  Baseline anxiety | 58.47 (5.39)
  Post-intervention anxiety: number analyzed (Participants) | 16
  Post-intervention anxiety | 57.49 (6.65)

7. Secondary Outcome: Patient-reported Stress
Description: Measured using using the Perceived Stress Scale (PSS-4), which assesses how overloaded, unpredictable, and uncontrollable respondents perceive their lives to be. The minimum score is 0 and the maximum score is 16, with higher scores indicating a higher stress level.
Time Frame: Measured at baseline (pre-intervention) and post-intervention (7-weeks).
Population: n=16 were retained at post-intervention
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Intervention
Number analyzed (Participants) | 33
Scores on a Scale
  Baseline stress | 5.55 (2.95)
  Post-intervention stress: number analyzed (Participants) | 16
  Post-intervention stress | 4.94 (4.11)

8. Secondary Outcome: Patient-reported Depression
Description: Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0 - Depression computer adaptive test which assesses self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Higher scores indicate higher levels of depression. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Measured at baseline (pre-intervention) and post-intervention (7-weeks).
Population: n=16 were retained at post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention
Number analyzed (Participants) | 33
T-score
  Baseline depression | 53.58 (5.72)
  Post-intervention depression: number analyzed (Participants) | 16
  Post-intervention depression | 52.52 (8.00)

9. Secondary Outcome: Patient-reported Positive Affect
Description: Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0- Positive Affect computer adaptive test, which assesses momentary positive or rewarding affective experiences, such as feelings and mood associated with pleasure, joy, elation, contentment, pride, affection, happiness, engagement, and excitement. Higher scores indicate higher levels of positive affect. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Measured at baseline (pre-intervention) and post-intervention (7-weeks).
Population: n=16 were retained at post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention
Number analyzed (Participants) | 33
T-score
  Baseline positive affect | 41.42 (6.65)
  Post-intervention positive affect: number analyzed (Participants) | 16
  Post-intervention positive affect | 42.31 (9.08)

10. Secondary Outcome: Patient-reported Meaning and Purpose
Description: Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0- Meaning and Purpose computer adaptive test, which assesses one's sense of life having purpose and that there are good reasons for living. Higher scores indicate hopefulness, optimism, goal-directedness, and feelings that one's life is worthy. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Measured at baseline (pre-intervention) and post-intervention (7-weeks).
Population: n=1 did not complete this measure at baseline; n=16 were retained at post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention
Number analyzed (Participants) | 32
T-score
  Baseline meaning and purpose | 45.51 (9.5)
  Post-intervention meaning and purpose: number analyzed (Participants) | 16
  Post-intervention meaning and purpose | 48.23 (11.74)

ADVERSE EVENTS:
Time Frame: from enrollment until post-intervention, 7 weeks
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

LIMITATIONS AND CAVEATS:
Given the small sample size, this study is not powered to detect statistically significant changes. This is a single-arm trial; therefore, any changes from baseline to post-intervention cannot necessarily be attributed to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT06359314/Prot_SAP_000.pdf